CLINICAL TRIAL: NCT04674787
Title: Uncertainty Analysis of Computational Model to Simulate Neurostimulation Caused by Gradient Fields in MRI
Acronym: NEUROMAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bryn Lloyd (Other)
Collaborators: Institute for Biomedical Engineering, Swiss Federal Institute of Technology (ETH Zurich) (Unknown)
Responsible Party: Sponsor-Investigator, Bryn Lloyd, Project Leader, The Foundation for Research on Information Technologies in Society (IT'IS), Switzerland
Organization: The Foundation for Research on Information Technologies in Society (IT'IS), Switzerland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: NEUROMAN
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Peripheral Nerve Stimulation in MRI; Electric Stimulation
Keywords: MRI gradient coil; peripheral nerve stimulation; Time varying magnetic fields

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Peripheral nerve stimulation provocation study — Study which measures stimulation thresholds in volunteers induced by low frequency electromagnetic gradients used in MRI scanners.

SUMMARY:
The aim of this research project is to quantify the uncertainty of current state-of-the art anatomical phantoms and computational models for predicting neurostimulation induced by time-varying magnetic fields (so-called gradient fields) within the context of magnetic resonance imaging (MRI) scanners. For this purpose stimulation thresholds will be measured in a volunteer study. The measurements will provide valuable data for the development and validation of future models.

DETAILED DESCRIPTION:
The study does not investigate any health related interventions, neither a therapy nor medical device. The study aims to provoke peripheral nerve stimulation from time varying magnetic (so-called "gradient") fields in volunteers in order to measure gradient threshold levels in different configurations (different gradient coil units, different positions and postures). The experiments will provide new data regarding the interaction of gradient fields and function of the peripheral nervous system. These measurements are of general interest to quantify associated modeling uncertainties and validate current or future computational modeling techniques.

The experiments will use an MR scanner to generate the gradient fields used to induce stimulation. In normal mode the maximum gradient field allowed by the manufacturer may lead to peripheral nerve stimulation in approximately 50% of subjects. However, depending on the position and posture it may induce PNS in even fewer than 50% of subjects. Therefore, for the purpose of measuring stimulation thresholds it is necessary to operate the gradient units in experimental mode (with respect to the gradient field) as described in IEC 60601-2-33, i.e. the gradient limits set by the manufacturer will be disabled. As described in the standard, the gradient field will be increased slowly from non-stimulating levels until the volunteer perceives first stimulation sensations, at which point the gradient field will be stopped. This protocol does not lead to an increased risk of cardiac muscle stimulation compared to the normal mode, but only an increased likelihood of PNS with non-painful sensations in the skin, e.g. tingling, twitching or poking. PNS is not considered a health concern. The radio-frequency (RF) field will remain switched off, i.e. there is no risk of heating (the scanner will not acquire images in this mode).

ELIGIBILITY:
Inclusion Criteria:

* healthy adult volunteers (six female and six male)

Exclusion Criteria:

* pregnant woman
* metallic implants or a history of neurological or cardiovascular diseases
* children and persons who are not able to follow the instructions will be excluded, due to a higher risk and lack of direct benefits from participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Measure PNS stimulation thresholds | The experimental procedure will be conducted during a single visit of approx. 90 minutes.
  The primary objective is to measure PNS stimulation thresholds in order to quantify the modeling uncertainty and reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- IT'IS Foundation, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Stimulation thresholds and stimulation locations will be recorded for each stimulation configuration (81 measurements with different subject position, posture, slew rates).
  This stimulation measurement data will be shared after publication of our findings in anonymized form to allow other researchers to validate their models with the data.
Supporting Information: Study Protocol
Time Frame: After publication of our findings in a peer reviewed journal
Access Criteria: Openly available to interested parties.